CLINICAL TRIAL: NCT04969250
Title: SARS-CoV-2 Vaccination Strategies in Previously Hospitalized and Recovered COVID-19 Patients
Brief Title: Vaccination for Recovered Inpatients With COVID-19 (VATICO)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: University of Minnesota (Other); International Network for Strategic Initiatives in Global HIV Trials (INSIGHT) (Network); University of Copenhagen (Other); Kirby Institute (Other Government); Washington D.C. Veterans Affairs Medical Center (U.S. Federal Agency); Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network); National Heart, Lung, and Blood Institute (NHLBI) (NIH); US Department of Veterans Affairs (U.S. Federal Agency); Prevention and Early Treatment of Acute Lung Injury (Other); Cardiothoracic Surgical Trials Network (Other); Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 016 / VATICO
Record Dates: First submitted 2021-07-16; First posted 2021-07-20 (Actual); Results first posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Covid19
Keywords: COVID-19; COVID 19; Coronaviridae Infections; Coronavirus Infections; RNA Virus Infections; Virus Diseases; Nidovirales Infections; SARS-CoV-2; SARS Coronavirus; VATICO; ACTIV-3; ACTIV3; TICO
MeSH Terms: conditions — COVID-19; Coronaviridae Infections; Coronavirus Infections; RNA Virus Infections; Virus Diseases; Nidovirales Infections; Severe Acute Respiratory Syndrome | interventions — 2019-nCoV Vaccine mRNA-1273; BNT162 Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Group I1 (Experimental): Immediate, one dose. Vaccination at study entry
  Interventions: Biological: Moderna mRNA-1273 COVID-19 vaccine; Biological: Pfizer BNT162b2 COVID-19 vaccine
- Group I2 (Experimental): Immediate, two doses. Vaccination at study entry and Week 4
  Interventions: Biological: Moderna mRNA-1273 COVID-19 vaccine; Biological: Pfizer BNT162b2 COVID-19 vaccine
- Group D1 (Experimental): Deferred, one dose. Vaccination at Week 12 only
  Interventions: Biological: Moderna mRNA-1273 COVID-19 vaccine; Biological: Pfizer BNT162b2 COVID-19 vaccine
- Group D2 (Experimental): Deferred, two doses. Vaccination at Week 12 and Week 16
  Interventions: Biological: Moderna mRNA-1273 COVID-19 vaccine; Biological: Pfizer BNT162b2 COVID-19 vaccine

INTERVENTIONS:
Biological: Moderna mRNA-1273 COVID-19 vaccine — 100 µg intramuscular injection
Biological: Pfizer BNT162b2 COVID-19 vaccine — 30 µg intramuscular injection

SUMMARY:
In this Phase 4, open-label trial, participants of the ACTIV-3/TICO clinical trial at selected sites who received certain pre-specified blinded investigational agents or placebo as part of that trial, and who have since achieved sustained recovery, and who are still [TICO assignment] blinded and who are still within 28 to 90 days after initial TICO randomization, will be randomized in this 2x2 factorial design to one of four groups: (i) immediate versus 12 week deferral of first dose administration and also (ii) one dose only, versus two doses to be given 4 weeks apart of the Moderna mRNA-1273 or the Pfizer BNT162b2 vaccine (mRNA vaccines).

Choice of Moderna or Pfizer vaccine is determined based on availability at the site. The choice is individual, although participants vaccinated twice should receive the same type of vaccine for both injections. The primary objectives of this 2x2 factorial design are (i) to estimate the difference in neutralizing antibody (NAb) response to the mRNA vaccine from baseline to Week 48 among participants vaccinated early versus deferred, and (ii) to estimate the difference in NAb response to this vaccine among participants vaccinated once versus twice. The primary analyses will be carried out in participants randomized to placebo in TICO. Analyses will also be carried out for those who receive the investigational agent(s) studied in TICO.

A key secondary objective is to ascertain the effect, if any, of SARS-CoV-2 monoclonal antibodies, and other interventions that have been studied in hospitalized COVID-19 subjects, on natural and vaccine-induced immunity.

Participants will remain blinded to the interventions received in the ACTIV-3/TICO study, however allocation to the timing of vaccination and to one or two vaccinations in this (VATICO) study is not blinded.

DETAILED DESCRIPTION:
In this Phase 4 trial, participants in the TICO master protocol who received certain pre-specified blinded investigational agents or matched placebos will be offered enrollment, with the understanding that this will require 2X2 randomized assignment of the timing and of the number of mRNA SARS-CoV-2 vaccinations to be received, via publicly-available mRNA SARS-CoV-2 vaccination sites or via other routes, in keeping with the 4 specified study arm assignments.

This will address the objective of evaluating if the vaccine is best administered early or deferred after recovery, and whether one injection provides comparable immune response to a two-injection course of vaccination. Participants (as well as the protocol team) will remain blinded to the interventions studied in TICO. Allocation to timing of vaccination and to one or two vaccinations is not blinded. Participants will be offered enrollment in this protocol at the Day 28 or Day 90 visits in TICO, or anytime between these visits.

Participants will have blood collected for research purposes at the time of enrollment and at Weeks 12, 24, and 48.

The study vaccine and regimen will not be blinded; there will be be no 'dummy/placebo' vaccine administered. Vaccines are expected to be made available either through the study directly, or through a reliable public vaccination program using vaccine available per the local regulatory mechanism (e.g., currently under Emergency Use Authorization (EUA) for the United States) or via other routes in case such local mechanisms are not available.

Participants will be equally allocated to 4 groups to inform each of two vaccine strategies:

* One injection versus two (for the immediate and deferred groups)
* Immediate versus deferred (for one and two vaccinations)

Hence, the outcome of the randomization will lead to one of the four following vaccination strategies for each study participant:

I1 - Immediate, one dose: vaccination at study entry only I2 - Immediate, two doses: vaccination at study entry and Week 4 D1 - Deferred, one dose: vaccination at Week 12 only D2 - Deferred, two doses: vaccination at Week 12 and Week 16

Randomization will be stratified by study site and by randomization assignment in TICO for certain pre-specified investigational agents or their matching placebo.

When addressing the two co-primary objectives, the following groups are combined:

* Immediate vs deferred vaccine: groups I1 and I2 versus D1 and D2
* One versus two vaccinations: groups I1 and D1 versus I2 and D2

Similar comparisons will be made separately for each of the two principal TICO arms, i.e., for those assigned to one of the investigational agents and for those assigned to the matching placebo. Both of these comparisons are protected by the randomization in the present study.

Given the factorial design, whether there is an interaction of one factor (timing of vaccination) with the other factor (number of doses) will need to be assessed although the study is not fully powered for this evaluation.

A key secondary objective is to address whether the investigational agent studied in TICO (versus matching placebo) is affecting the primary outcome in this protocol. Of note, this comparison may not always be protected by randomization, as there may be differential inclusion in this protocol between those receiving the investigational agent in TICO and those receiving its matching placebo. This is more likely to be the case if the investigational agent is demonstrated to affect the chance of achieving sustained recovery.

The primary endpoint, immune response specific to the vaccination received, will be assessed at Week 48. Participants will have blood collected at time of enrollment, and at Weeks 12, 24 and 48 after study entry. Approximately 640 participants will be recruited. The total sample size will depend on how many investigational agents/placebo are evaluated in ACTIV-3/TICO.

ELIGIBILITY:
Inclusion Criteria:

* Participating in the ACTIV-3/TICO trial and received a selected blinded investigational agent, or placebo for that agent, at selected sites.
* Willingness to strictly adhere to the randomly allocated dosage number and schedule for vaccine administration.
* Participant is between Day 28 and Day 90 TICO visits inclusive at time of randomization.
* At time of screening for this study, has experienced sustained recovery (i.e., the primary endpoint in TICO) for at least two consecutive weeks, i.e. having returned uninterrupted to the person's premorbid living facility (or equivalent) for at least 2 consecutive weeks.
* Ability and willingness of participant (or legally authorized representative) to provide informed consent prior to initiation of any study procedures.

Exclusion Criteria:

* Receipt of a SARS-CoV-2 (COVID-19) vaccine after enrollment into TICO. Participants who received a SARS-CoV-2 vaccine prior to enrollment in TICO may be enrolled in this study.
* Known allergy to any component of the study eligible vaccine(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-08-25 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2022-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Jens Lundgren, Principal Investigator — INSIGHT Copenhagen International Coordinating Centre, Rigshospitalet, University of Copenhagen
Locations (30):
- United States (16):
  - Cedars-Sinai Medical Center (Site 208-002), 8700 Beverly Blvd, Los Angeles, California
  - San Francisco VAMC (Site 074-002), 4150 Clement Street, San Francisco, California
  - Stanford University Hospitals & Clinics (Site 203-003), Stanford University, School of Medicine, 300 Pasteur Dr., Grant Bldg, Room S011, Stanford, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Site 066-002), 1124 W. Carson St., CDCRC, Torrance, California
  - Public Health Institute at Denver Health (Site 017-004), 660 Bannock Street, Denver, Colorado
  - Washington DC VA Medical Center (Site 009-004), 50 Irving Street, NW., Washington D.C., District of Columbia
  - Hillsborough County Health Department, University of South Florida (Site 032-001), 1105 E. Kennedy Blvd., Tampa, Florida
  - Minneapolis VA Medical Center (Site 105-001), 1 Veterans Drive, Minneapolis, Minnesota
  - Duke University Hospital (Site 301-006), 2301 Erwin Road, Durham, North Carolina
  - Wake Forest Baptist Health (Site 210-001), Medical Center Boulevard, Winston-Salem, North Carolina
  - Rhode Island Hospital (Site 080-036), 593 Eddy St., Providence, Rhode Island
  - The Miriam Hospital (Site 080-039), 164 Summit Ave., Providence, Rhode Island
  - CHRISTUS Spohn Shoreline Hospital (Site 080-001), 600 Elizabeth Street, Corpus Christi, Texas
  - UT Southwestern Medical Center (Site 084-001), 1936 Amelia Court, 2nd Floor, Dallas, Texas
  - Parkland Health and Hospital Systems (Site 084-002), James Aston Ambulatory Care Center - Clinical Research Unit, 5303 Harry Hines Blvd., Ste U-9.300, Dallas, Texas
  - Salem VA Medical Center (Site 074-014), 1970 Roanoke Blvd., Salem, Virginia
- Institute of Human Virology-Nigeria (Site 612-601), International Research Center of Excellence, Cadastral Zone COO Plot 62, after BAZE University, off CITEC Road, Abuja, Nigeria
- Tan Tock Seng Hospital (Site 612-201), National Center for Infectious Diseases (NCID), 11 Jalan Tan Tock Seng, Singapore, Singapore
- Spain (5):
  - Hospital Universitari Vall d'Hebron (Site 626-033), Passeig Vall Hebron, 119-129, Barcelona
  - Hospital Clinic de Barcelona (Site 626-004), Carrer de Villaroel 170, Barcelona
  - Hospital Universitari Germans Trias i Pujol (Site 626-003) Carretera de Canyet, s/n, Barcelona
  - Hospital Universitari Arnau de Vilanova (Site 026-035), Institut de Recerca Biomèdica de Lleida, Av. Rovira Roure, 80, Lleida
  - Hospital General Universitario Gregorio Marañón (Site 626-001), Servicio de Inmunología Clínica, Departamento de Medicina Interna, Dr. Esquerdo, 46, Madrid
- University Hospital Zurich (Site 621-201), Raemistrasse 100, Zurich, Switzerland
- Uganda (6):
  - MRC/UVRI & LSHTM Uganda Research Unit (Site 634-601), Plot 51-59 Nakiwogo Road, P.O. Box 49, Entebbe
  - Gulu Regional Referral Hospital (Site 634-603), P.O. Box 160, Gulu
  - St. Francis Hospital, Nsambya (Site 634-607), Nsambya Road Nsambya Hill, P.O. Box 7146, Kampala
  - Makerere University Lung Institute (634-604), Mulago National Referral Hospital, Kampala
  - Lira Regional Referral Hospital (Site 634-605), Plot 9/19, 21-41 Ngetta Road Police Road, Lira
  - Masaka Regional Referral Hospital (Site 634-606), MRC/UVRI and LSHTM Uganda Research Unit, Plot 6 Circle Road, PO Box 556, Masaka

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: CDC (Centers for Disease Control and Prevention): Coronavirus (COVID-19) website — https://www.cdc.gov/coronavirus/2019-nCoV/index.html
- See also: A Participant's Guide to Clinical Trials (NIAID) — https://www.niaid.nih.gov/clinical-trials/participant-guide
- See also: Find a Clinical Trial — https://www.niaid.nih.gov/clinical-trials/find-a-clinical-trial
- See also: Clinical Trials at NIAID — https://www.niaid.nih.gov/clinical-trials
- See also: National Institute for Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: WHO COVID-19 treatment guidelines — https://www.who.int/emergencies/diseases/novel-coronavirus-2019/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The number of participants consented was not collected, so these numbers are the number of participants randomized.
Period: Overall Study
Arm/Group | Group I1 | Group I2 | Group D1 | Group D2
Started | 16 | 18 | 16 | 16
Completed | 16 | 15 | 13 | 8
Not Completed | 0 | 3 | 3 | 8
Not completed — Protocol Violation | 0 | 2 | 3 | 8
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I1 | Group I2 | Group D1 | Group D2 | Total
Number analyzed (Participants) | 16 | 18 | 16 | 16 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 15 | 13 | 15 | 55
  >=65 years | 4 | 3 | 3 | 1 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 6 | 8 | 28
  Male | 8 | 12 | 10 | 8 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 3 | 3 | 13
  Not Hispanic or Latino | 13 | 14 | 13 | 13 | 53
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 8 | 8 | 7 | 9 | 32
  White | 5 | 5 | 5 | 4 | 19
  More than one race | 0 | 1 | 2 | 1 | 4
  Other | 0 | 1 | 0 | 0 | 1
  Only ethnicity reported | 3 | 3 | 1 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Ratio of 48-Week to Baseline Neutralizing Antibody (NAb) Levels
Description: Change in antibody level as measured by ratio of follow-up to baseline level
Time Frame: Pre-vaccination baseline and 48 weeks post-vaccination
Population: Patient counts for this analysis are less than the total number of patients followed because some patients with follow-up visits did not have blood drawn.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio of geometric mean responses
Arm/Group | Group I1 | Group I2 | Group D1 | Group D2
Number analyzed (Participants) | 12 | 15 | 13 | 11
ratio of geometric mean responses | 0.3722 [-0.0566 to 0.8012] | 0.5883 [0.1366 to 1.0399] | 0.2088 [-0.1758 to 0.5935] | 0.3073 [-0.1479 to 0.7624]

2. Secondary Outcome: Ratio of 12-Week to Baseline Neutralizing Antibody (NAb) Levels
Description: Change in antibody level as measured by ratio of follow-up to baseline level
Time Frame: Pre-vaccination baseline and 12 weeks post-vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio of geometric mean responses
Arm/Group | Group I1 | Group I2 | Group D1 | Group D2
Number analyzed (Participants) | 13 | 15 | 14 | 13
Ratio of geometric mean responses | 0.4827 [0.0641 to 0.9014] | 0.9206 [0.4938 to 1.3474] | 0.2418 [-0.1329 to 0.6165] | 0.6533 [0.1554 to 1.1513]

3. Secondary Outcome: Ratio of 24-Week to Baseline Neutralizing Antibody (NAb) Levels
Description: Change in antibody level as measured by ratio of follow-up to baseline level
Time Frame: Pre-vaccination baseline and 24 weeks post-vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio of geometric mean responses
Arm/Group | Group I1 | Group I2 | Group D1 | Group D2
Number analyzed (Participants) | 14 | 16 | 14 | 12
Ratio of geometric mean responses | 0.3002 [-0.0453 to 0.6458] | 0.7747 [0.4187 to 1.1306] | 0.2032 [-0.1265 to 0.5328] | 0.3397 [-0.0498 to 0.7292]

4. Secondary Outcome: Number of Deaths
Description: Count of Deaths
Time Frame: Through Week 24 after enrollment
Population: Participant who withdrew consent was not included in analysis. Used Fisher's exact test rather than Chi-squared due to small N.
Measure: Count of Participants; unit: Participants
Arm/Group | Group I1 | Group I2 | Group D1 | Group D2
Number analyzed (Participants) | 16 | 17 | 16 | 16
Participants | 1 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Group I1 vs Group I2 vs Group D1 vs Group D2; Test type: Superiority; p = 0.73, Fisher Exact

5. Secondary Outcome: Number of Serious Adverse Events (SAEs)
Description: Count of SAEs
Time Frame: Through Week 24
Population: as for outcome 4
Measure: Number; unit: SAEs
Arm/Group | Group I1 | Group I2 | Group D1 | Group D2
Number analyzed (Participants) | 16 | 17 | 16 | 16
SAEs | 2 | 0 | 0 | 1
Statistical Analysis 1: Comparison: Group I1 vs Group I2 vs Group D1 vs Group D2; Test type: Superiority; p = 0.40, Fisher Exact

6. Secondary Outcome: Number of Patients Non-adherent to 2nd Dose
Description: Number of participants assigned a 2nd vaccine dose who did not receive it for any reason
Time Frame: Second vaccine doses were due at 4 and 16 weeks after randomization in Arm 2 and 4, respectively
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Group I2 | Group D2
Number analyzed (Participants) | 17 | 16
Participants | 1 | 5
Statistical Analysis 1: Comparison: Group I2 vs Group D2; Test type: Superiority; p = 0.078, Fisher Exact

7. Secondary Outcome: Number of Patients Non-adherent to Assigned Treatment Strategy
Description: Number of participants who received more or less vaccine than assigned, or who received vaccines at different time points than assigned
Time Frame: Vaccine doses were due through 16-weeks post-randomization; participants were followed for vaccination status through 48 weeks post-randomization
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Group I1 | Group I2 | Group D1 | Group D2
Number analyzed (Participants) | 16 | 17 | 16 | 16
Participants | 1 | 3 | 5 | 8
Statistical Analysis 1: Comparison: Group I1 vs Group I2 vs Group D1 vs Group D2; Test type: Superiority; p = 0.033, Fisher Exact

8. Secondary Outcome: Percent of Patients With >=4-fold Difference in NAb
Description: Percentage of participants with >=4-fold change in NAb from baseline to 48 weeks
Time Frame: Pre-vaccination baseline and 48 weeks post-vaccination
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Group I1 | Group I2 | Group D1 | Group D2
Number analyzed (Participants) | 12 | 15 | 13 | 11
percentage of participants | 41.70 | 53.30 | 30.80 | 27.30

ADVERSE EVENTS:
Time Frame: 48 weeks
Description: Participant who withdrew consent was not included in analysis.
Arm/Group | Group I1 | Group I2 | Group D1 | Group D2
All-Cause Mortality (participants affected / at risk) | 1/16 | 0/17 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 1/16 | 0/17 | 0/16 | 1/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/17 | 0/16 | 0/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I1 (N=16) | Group I2 (N=17) | Group D1 (N=16) | Group D2 (N=16)
Acute chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aggravation of bicytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Recurrence of COVID-19 infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This trial anticipated enrolling 640 participants, but enrolled just 66.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol: Protocol (2021-06-07): https://cdn.clinicaltrials.gov/large-docs/50/NCT04969250/Prot_000.pdf
  • Study Protocol: Letter of Amendment (2021-08-03): https://cdn.clinicaltrials.gov/large-docs/50/NCT04969250/Prot_001.pdf
  • Statistical Analysis Plan (2023-08-31): https://cdn.clinicaltrials.gov/large-docs/50/NCT04969250/SAP_004.pdf
  • Informed Consent Form (2021-08-03): https://cdn.clinicaltrials.gov/large-docs/50/NCT04969250/ICF_003.pdf